CLINICAL TRIAL: NCT01233232
Title: A 4 Week, Double Blind, Placebo Controlled, Randomised, Parallel Group, Multicentre, Phase IIa Study to Investigate the Safety and Tolerability of AZD5069 as Oral Capsules in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A 4 Week Study to Investigate the Safety and Tolerability of AZD5069 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Acronym: CIRRUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3550C00002; 2010-021217-23 (EudraCT Number)
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-08

CONDITIONS: Scientific Terminology Chronic Obstructive Pulmonary Disease (COPD); Laymen Terminology Chronic Bronchitis and Emphysema
Keywords: Chronic Obstructive Pulmonary Disease, Neutrophil, Respiratory Disease
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Respiration Disorders | interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Placebo Comparator): Placebo dose
  Interventions: Drug: Placebo
- 2 (Experimental): Treatment arm AZD5069 50mg
  Interventions: Drug: AZD5069 50mg
- 3 (Experimental): Treatment arm AZD5069 80mg
  Interventions: Drug: AZD5069 80mg

INTERVENTIONS:
Drug: Placebo — Oral dose bid
  Arms: 1
Drug: AZD5069 50mg — Oral dose bid
  Arms: 2
Drug: AZD5069 80mg — Oral dose bid
  Arms: 3

SUMMARY:
The purpose of this study is the evaluate the safety and tolerability of AZD5069 in patients with Chronic Obstructive Pulmonary Disease

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD with symptoms for more than one year before screening
* Body mass index of 18-30 kg/m2 and weight of 50-100kg
* Current or ex-smokers with a smoking history of at least 10 pack years (1 pack year = tobacco consumption corresponding to 20 cigarettes smoked per day for one year) at screening
* FEV1 of 30% or above and less than 80% of the predicted normal value post-bronchodilator at screening
* FEV1/FVC less than 70% post-bronchodilator at screening

Exclusion Criteria:

* Any clinically significant disease or disorder
* Exacerbation of COPD which was not resolved within 30 days of first dosing
* Patients who have received live or live-attenuated vaccine in the 2 weeks prior to first dosing
* Asthma and any current respiratory tract disorder other than COPD which is considered to be clinically significant
* Disease history suggesting reduced or abnormal immune function other than that related to COPD

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Research Site, Sofia, Bulgaria
- Germany (2):
  - Research Site, Berlin
  - Research Site, Großhansdorf
- Hungary (4):
  - Research Site, Debrecen
  - Research Site, Pécs
  - Research Site, Százhalombatta
  - Research Site, Szeged
- Research Site, Kyiv, Ukraine

REFERENCES:
- [Background] Kirsten AM, Forster K, Radeczky E, Linnhoff A, Balint B, Watz H, Wray H, Salkeld L, Cullberg M, Larsson B. The safety and tolerability of oral AZD5069, a selective CXCR2 antagonist, in patients with moderate-to-severe COPD. Pulm Pharmacol Ther. 2015 Apr;31:36-41. doi: 10.1016/j.pupt.2015.02.001. Epub 2015 Feb 11. PMID 25681277
- See also: D3550C00002_Revised_Clinical_Study_Protocol.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=208&filename=D3550C00002_Revised_Clinical_Study_Protocol.pdf
- See also: D3550C00002_Study_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=208&filename=D3550C00002_Study_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 22 November 2010. Last patient completed: 22 March 2011. Fifteen centres across 4 countries participated in this study: Bulgaria (4), Germany (4), Hungary (4) and Ukraine (3)
Pre-assignment Details: 22 patients enrolled were not randomized due to eligibility not fulfilled (17 patients) and voluntary discontinuation (5 patients)
Groups:
- Placebo: 4 x placebo capsules, twice daily (bid)
- AZD5069 50 mg: 1 x 50 mg AZD5069 capsule and 3 x placebo capsules, bid
- AZD5069 80 mg: 4 x 20 AZD5069 mg capsules, bid
Period: Overall Study
Arm/Group | Placebo | AZD5069 50 mg | AZD5069 80 mg
Started | 29 | 30 | 28
Completed | 28 | 30 | 28
Not Completed | 1 | 0 | 0
Not completed — Voluntary Discontinuation by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AZD5069 50 mg | AZD5069 80 mg | Total
Number analyzed (Participants) | 29 | 30 | 28 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (7.9) | 65 (6.9) | 65 (7.4) | 64 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 6 | 27
  Male | 20 | 18 | 22 | 60
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.842 (2.77) | 27.645 (2.89) | 25.803 (3.18) | 26.118 (3.14)
Weight [Mean (Standard Deviation); unit: Kg] | 73.7 (14.02) | 78.9 (9.18) | 75.4 (10.90) | 76 (11.59)
% Predicted FEV1 at screening [Mean (Standard Deviation); unit: %] | 56 (13.9) | 57 (13.6) | 54 (12.1) | 56 (13.2)
FEV1/FVC at screening [Mean (Standard Deviation); unit: %] | 52.54 (9.62) | 51.75 (11.65) | 54.52 (10.51) | 52.91 (10.58)
Nicotine pack years [Mean (Standard Deviation); unit: Pack Year] — one pack year= 1 pack (20 cigrettes) per day for 1 year, or equivalent
  Pack Year | 38 (21.4) | 39 (22) | 34 (17.9) | 37 (20.4)
GOLD classification [Number; unit: Participants] — The spirometric classification of severity COPD now includes four stages: Stage I: Mild; Stage II: Moderate; Stage III: Severe; Stage IV: Very Severe.
  Participants
    II Moderate | 17 | 20 | 16 | 53
    III Severe | 12 | 10 | 12 | 34

OUTCOME MEASURES:

1. Primary Outcome: Patients Who Experienced at Least One Adverse Events(s)
Description: Adverse event (AE) data, both serious and non-serious. An AE is the development of an undesirable medical condition (eg, nausea, chest pain, tachycardia, laboratory findings) or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.
Time Frame: From start of treatment (Day 0) up to 28 days (End of Treatment)
Measure: Number; unit: Participants
Groups:
- Arm 1 - Placebo: 4 x placebo capsules, twice daily (bid)
- Arm 2 - AZD5069 50 mg: 1 x 50 mg AZD5069 capsule and 3 x placebo capsules, bid
- Arm 3 - AZD5069 80 mg: 4 x 20 AZD5069 mg capsules, bid
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 29 | 30 | 28
Participants | 9 | 10 | 6

2. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination includes assessment of general appearance, skin, head and neck (including ears, eyes, nose and throat), lymph nodes, musculo-skeletal (including spine and extremities), cardiovascular, lungs and abdomen. The findings were deemed to be normal/abnormal based on the clinical judgment of the investigator.
Time Frame: Last Observation on Treatment (up to Day 28)
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 29 | 30 | 28
Participants | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG)
Description: ECGs were recorded in the supine position after the patient has rested for 10 minutes. Heart rate, QRS duration, PR, RR and QT intervals were recorded. Overall evaluation of the ECG is classified as normal, abnormal or borderline. Only participants with ECG at baseline classified as normal are reported (ie, only changes from normal to abnormal).
Time Frame: Baseline (last non-missing assessment prior to first dose of study medication) and End of Treatment (Day 28)
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 22 | 25 | 23
Participants | 0 | 0 | 0

4. Primary Outcome: Change From Baseline to End of Treatment for Leucocytes Count in Blood (Safety Blood Sample)
Description: The change in circulating leucocyte counts (including neutrophils) is calculated as the End of Treatment value minus the Baseline value.
Time Frame: Baseline (last non-missing assessment prior to first dose of study medication) and End of Treatment (Day 28)
Measure: Mean (Standard Deviation); unit: 10^9/L cells/L
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 28 | 28 | 28
10^9/L cells/L | -0.12 (1.974) | -1.55 (2.059) | -1.08 (2.404)

5. Primary Outcome: Change From Baseline to End of Treatment for Body Temperature
Description: The change in body temperature (oral) is calculated as the End of Treatment value minus the Baseline value.
Time Frame: Baseline (last non-missing assessment prior to first dose of study medication) and End of Treatment (Day 28)
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 28 | 30 | 28
degrees C | -0.1 (0.43) | 0.0 (0.57) | -0.0 (0.39)

6. Primary Outcome: Change From Baseline to End of Treatment for Systolic Blood Preassure (Vital Signs)
Description: The change in systolic blood pressure (Vital Sign) is calculated as the End of Treatment value minus the Baseline value.
Time Frame: Baseline (last non-missing assessment prior to first dose of study medication) and End of Treatment (Day 28)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 28 | 30 | 28
mmHg | 3.0 (11.0) | -0.0 (12.1) | -3.0 (15.7)

7. Primary Outcome: Change From Baseline to End of Treatment for Diastolic Blood Pressure (Vital Signs)
Description: The change in diastolic blood pressure (Vital Sign) is calculated as the End of Treatment value minus the Baseline value.
Time Frame: Baseline (last non-missing assessment prior to first dose of study medication) and End of Treatment (Day 28)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 28 | 30 | 28
mmHg | 2.0 (7.2) | -2.0 (7.9) | -1.0 (8.2)

8. Primary Outcome: Change From Baseline to End of Treatment for Pulse Rate (Vital Signs)
Description: The change in pulse rate (Vital Sign) is calculated as the End of Treatment value minus the Baseline value.
Time Frame: Baseline (last non-missing assessment prior to first dose of study medication) and End of Treatment (Day 28)
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 28 | 30 | 28
beats/minute | 1 (6.2) | -1 (6.9) | 3 (7.9)

9. Primary Outcome: Change From Baseline to End of Treatment for FEV1 Pre-bronchodilator (Lung Function Test)
Description: The change in FEV1 Pre-bronchodilator is calculated as the End of Treatment value minus the Baseline value.
Time Frame: Baseline (last non-missing assessment prior to first dose of study medication) and End of Treatment (Day 28)
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 28 | 30 | 27
L | -0.03 (0.238) | 0.05 (0.238) | -0.01 (0.218)

10. Primary Outcome: Change From Baseline to End of Treatment for FEV1 Post-bronchodilator (Lung Function Test)
Description: The change in FEV1 Post-bronchodilator is calculated as the End of Treatment value minus the Baseline value.
Time Frame: Baseline (last non-missing assessment prior to first dose of study medication) and End of Treatment (Day 28)
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 27 | 30 | 28
L | -0.02 (0.230) | 0.10 (0.256) | 0.02 (0.194)

11. Primary Outcome: Number of Participants Who Developed High Transaminase Values (Clinical Chemistry)
Description: High Transaminase Values are defined as a measurment of ALT (alanine aminotransferase) or AST (aspartate aminotransferase) greater than or equal to 3 times the upper limit of normal (ALT ULN = 36 IU/L, AST ULN = 33 IU/L).
Time Frame: Up to Follow-up Visit (3 to 18 days after End of Treatment [Day 28])
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 29 | 30 | 28
Participants | 0 | 0 | 0

12. Primary Outcome: Change From Baseline to End of Treatment for Total Protein (Urinalysis)
Description: The change in total protein in urine is calculated as the End of Treatment value minus the Baseline value.
Time Frame: Baseline (last non-missing assessment prior to first dose of study medication) and End of Treatment (Day 28)
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 6 | 4 | 1
g/L | -0.02 (0.034) | -0.01 (0.022) | -0.01 (NA) — Only one value in arm 3. SD is not calculable.

13. Secondary Outcome: Plasma Concentration of AZD5069 After 1 Hour of Dosing
Description: At this visit, approximately 1 hour after dosing (at the clinic), a blood sample was collected for determination of drug concentration in plasma.
Time Frame: End of Treatment (Day 28), 1 hour after dosing
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 0 | 18 | 18
nmol/L |  | 2599.551 (2085.601) | 5433.611 (4622.932)

14. Secondary Outcome: Area Under the Plasma Concentration Curve of AZD5069
Description: The area under the plasma concentration curve is estimated from time 0 (dosing) to 24 hours after dosing.
Time Frame: End of Treatment (Day 28); pre-dose, 1, 2, 3, and 5 hours after dosing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 26 | 22
nmol*h/L | 29600 (108) [4270 to 136000] | 38800 (95.6) [6700 to 143000]

15. Secondary Outcome: Maximum Plasma Concentration for AZD5069
Description: The maximum plasma concentration (Cmax) is the highest level of drug in plasma.
Time Frame: End of Treatment (Day 28); pre-dose, 1, 2, 3, and 5 hours after dosing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 26 | 22
nmol/L | 2550 (107) [367 to 11700] | 3340 (95.6) [576 to 12300]

16. Secondary Outcome: Time to Maximum Plasma Concentration for AZD5069
Description: Time (in relation to dosing) at which the maximum plasma concentration is observed.
Time Frame: End of Treatment (Day 28); pre-dose, 1, 2, 3, and 5 hours after dosing
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 26 | 22
hours | 1.56 [1.56 to 1.56] | 1.56 [1.56 to 1.56]

17. Secondary Outcome: Maximum Reduction of Circulating Neutrophils in Blood, From Baseline
Description: The change in circulating neutrophils in blood is calculated as the visit value minus the Baseline value. Only participants with reduction are considered.
Time Frame: Baseline (last non-missing assessment prior to first dose of study medication), weeks 1, 2 and 3, and End of Treatment (Day 28)
Measure: Mean (Standard Deviation); unit: 10^9/L cells/L
Arm/Group | Arm 1 - Placebo | Arm 2 - AZD5069 50 mg | Arm 3 - AZD5069 80 mg
Number analyzed (Participants) | 22 | 30 | 26
10^9/L cells/L | 1.324 (1.2152) | 2.759 (1.4422) | 2.678 (2.0710)

ADVERSE EVENTS:
Arm/Group | Placebo | AZD5069 50 mg | AZD5069 80 mg
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/30 | 1/28
Other Adverse Events (participants affected / at risk) | 3/29 | 8/30 | 1/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | AZD5069 50 mg (N=30) | AZD5069 80 mg (N=28)
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | AZD5069 50 mg (N=30) | AZD5069 80 mg (N=28)
Nasopharyngitis (Infections and infestations) | 2 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Pyrexia (General disorders) | 2 | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 3 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less